CLINICAL TRIAL: NCT06013033
Title: DDX17 Orchestrate Septic Vascular Endothelial Pyroptosis by Controlling Gasdermin D Pore Formation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Fei Peng, Principal Investigator, Zhongda Hospital
Other Study IDs: 82202393
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3 mL of the patient's peripheral blood were drawn on Day1, 3, and 7, and the plasma was centrifuged and kept at -80 °C. ELISA content detection of DDX17 and GSDMD.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective: To investigate the correlation between plasma levels of DDX17 and GSDMD with vascular endothelial dysfunction and prognosis of in sepsis patients.

Design: A single center, prospective, observational research. Participants: Patients with sepsis who are hospitalized to Southeast University Affiliated Zhongda Hospital and meet the diagnostic criteria for sepsis 3.0.

Inclusion criteria:1. There is a potential or clear infection; 2. Sequential organ failure score (SOFA score) increases by more than or equal to 2 points compared to the baseline value; 3. Sign informed consent form.

Exclusion criteria: Age<18 years old or>80 years old, pregnant women, tumor patients, including diseases that may be complicated with vascular endothelial damage: hypertension, acute and chronic hepatitis (hepatitis caused by virus), liver cirrhosis, PT prolongation after liver transplantation, acute myocardial infarction, chronic tubular nephritis, chronic renal insufficiency/maintenance hemodialysis, renal transplantation, interstitial pneumonia, acute pancreatitis, active phase of systemic lupus erythematosus Ulcerative colitis, Crohn's disease, HELLP syndrome.

Primary outcome: 28-day mortality. Secondary outcome: Plasma levels of DDX17 and GSDMD, and their correlation with vascular endothelial injury, severity, and prognosis in sepsis patients.

DETAILED DESCRIPTION:
Data collection:Recording the population information, including name, sex, BMI, and past history. Recording disease-related information's, including diagnosis, infection site, pathogens, organ dysfunction, SOFA and APACHE II scores. Recording treatment measures of patients, including whether to use vasopressor, invasive mechanical ventilation, and continuous renal replacement therapy. Recording laboratory examination results, including leukocyte count, PCT and hs-CRP on D1, D3 and D7, respectively. All patients were followed up to 28 days. Patients were distributed to survival group and non-survival group according to the 28-day survival.

Sample collection: 3 mL of the patient's peripheral blood were drawn on Day1, 3, and 7, and the plasma was centrifuged and kept at -80 °C. ELISA content detection of DDX17 and GSDMD.

ELIGIBILITY:
Inclusion Criteria:

* There is a potential or clear infection;
* Sequential organ failure score (SOFA score) increases by more than or equal to 2 points compared to the baseline value;
* Sign informed consent form.

Exclusion Criteria:

* Age<18 years old or>80 years old
* pregnant women
* tumor patients
* including diseases that may be complicated with vascular endothelial damage: hypertension, acute and chronic hepatitis (hepatitis caused by virus), liver cirrhosis, PT prolongation after liver transplantation, acute myocardial infarction, chronic tubular nephritis, chronic renal insufficiency/maintenance hemodialysis, renal transplantation, interstitial pneumonia, acute pancreatitis, active phase of systemic lupus erythematosus Ulcerative colitis, Crohn's disease, HELLP syndrome.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis who are hospitalized to Southeast University Affiliated Zhongda Hospital and meet the diagnostic criteria for sepsis 3.0.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days

SECONDARY OUTCOMES:
correlation between plasma level of DDX17 and vascular endothelial injury, severity, and prognosis in sepsis patients | 28 days
correlation between plasma level of GSDMD and vascular endothelial injury, severity, and prognosis in sepsis patients | 28 days